CLINICAL TRIAL: NCT06398795
Title: Dual-port Trans-subclavian Thyroid Endoscopic Surgery - an Exploration of Cavity Construction in Situ Heralds a New Approach Choice
Brief Title: Dual-port Trans-subclavian Thyroid Endoscopic Surgery
Acronym: DTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YLJS-2022036-01
Record Dates: First submitted 2024-04-22; First posted 2024-05-03 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Neoplasms; Endoscopic Surgery
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTS group (Experimental): Patients undergo Dual-port Trans-subclavian Thyroid Endoscopic Surgery (DTS)
  Interventions: Procedure: Dual-port Trans-subclavian Thyroid Endoscopic Surgery (DTS).
- COT group (Active Comparator): Patients undergo conventional open thyroidectomy (COT)
  Interventions: Procedure: Conventional open thyroidectomy (COT)

INTERVENTIONS:
Procedure: Dual-port Trans-subclavian Thyroid Endoscopic Surgery (DTS). — An innovative surgical approach, Dual-port Trans-subclavian Thyroid Endoscopic Surgery (DTS), presents a unique dual-port endoscopic technique for thyroidectomy. DTS significantly reduces postoperative hospital stay, emphasizing its potential for accelerated patient recovery compared to COT.
  Arms: DTS group
Procedure: Conventional open thyroidectomy (COT) — open thyroidectomy with traditional collar incisions
  Arms: COT group

SUMMARY:
This is a prospective, single-center, open-label, non-randomized controlled real-world study aimed at exploring a novel approach to cavity construction for thyroid endoscopic surgery. The study seeks to evaluate its effectiveness and safety while accumulating further evidence-based medical data.

Three hundred patients with thyroid tumors were divided into an experimental group (150 cases receiving a new endoscopic thyroid surgery technique, namely, dual-port trans-subclavian thyroid endoscopic surgery) and a control group (150 cases undergoing traditional open thyroid surgery) according to their treatment intention. Laboratory and medical data from specified follow-up points are collected, and adverse events are recorded detailly.

The primary efficacy endpoint is a comparison of surgical complications between the two treatment groups. Secondary endpoints include: (1) levels of IL-2, IL-4, IL-6, IL-10, TNF-α, INF-γ, renin, angiotensin II, and aldosterone preoperatively and on the second day postoperatively; (2) NRS scores on the first day postoperatively; (3) length of hospital stay, duration of surgery, total treatment cost, and postoperative drainage volume; and (4) assessment of wound satisfaction during a three-month follow-up visit.

Safety assessments include adverse events, vital signs, and pathological examinations.

DETAILED DESCRIPTION:
In the past years, the prevalence of thyroid cancer (TC) has increased markedly across numerous regions and nations. 94% of TC are differentiated thyroid carcinomas (DTC), and thyroidectomyis widely accepted as the most optimal therapeutic option for patients diagnosed with DTC. The conventional method for performing thyroidectomy is through an open approach known as collar incision thyroidectomy, or conventional open thyroidectomy (COT), which is commonly recognized as the standard technique.

Endoscopic thyroid surgery is a relatively new approach to thyroid surgery that was first developed in the 1990s. In 1996, Dr. Hiischer, an Italian surgeon, performed the first endoscopic right thyroid lobectomy. Recently, with the advent of intraoperative neuromonitoring (IONM), a technique for monitoring recurrent laryngeal nerve (RLN) function during surgery, complications of RLN injury have been effectively reduced. The introduction of high-definition endoscopy and robotic surgery in endoscopic thyroid procedures has significantly enhanced visual precision, enabling surgeons to perform complex maneuvers with increased accuracy, thereby minimizing the risk of complications and tissue injury. With the advancement of these technologies, various endoscopic thyroidectomy techniques have been developed, including chest-breast, transoral, and transaxillary approaches.

However, in comparison to COT, endoscopic thyroid surgery incurs greater trauma. This is primarily attributed to the absence of initial spaces in the neck, unlike the thoracic and abdominal cavities. Previous endoscopic procedures required creating a cavity from a distance before extending it to the neck, leading to a direct increase in the surgical trauma area. Consequently, patients undergoing endoscopic thyroid surgery may endure more substantial surgical trauma, exacerbated postoperative pain, and prolonged hospitalization. Hence, some scholars argue that the transformation of endoscopic thyroid surgery into a genuinely 'minimally invasive procedure'; necessitates further refinement.

To address the aforementioned issue, the investigators propose a pioneering approach: Dual-port Trans-subclavian Thyroid Endoscopic Surgery (DTS) . DTS has the following advantages: 1) The investigators employed two 1cm puncture holes, thereby reducing the incision-related trauma to the skin and subcutaneous tissues, significantly alleviating surgical trauma and postoperative pain in patients. 2) The previous endoscopic approach involves creating an additional cavity, leading to additional trauma, whereas our method is directly constructing the cavity in situ within the neck. 3) Our endoscopic visual field is well-exposed, ensuring thorough clearance of central compartment lymph node.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid cancer or benign thyroid tumors
* Patients with a demand for incisional cosmetic improvement

Exclusion Criteria:

* Patients with thyroid cancer larger than 2 cm
* benign tumors larger than 5 cm
* Patients with severe underlying diseases
* Patients with chronic kidney disease,
* Patients with autoimmune diseases
* Patients with rheumatoid arthritis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative complications | From the date of grouping to the first recorded progression of relapse or the date of death due to any cause, whichever came first, assessed up to 100 months.
  The incidence of postoperative complications including recurrent laryngeal nerve injury, hypoparathyroidism, chyle leakage, infection and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jiashu Wu, Profe, Principal Investigator — The first hospital of Wenzhou Medical University
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No